CLINICAL TRIAL: NCT05602701
Title: Preoperative Prediction of Postoperative Physical Function in Patients With Total Knee Arthroplasty Based on Physical Fitness and Patient Characteristics: A Prospective Cohort Study
Brief Title: Preoperative Prediction of Postoperative Physical Function
Status: Terminated | Type: Observational
Why Stopped: Intended inclusion rate was not met
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Annadal Clinic (Unknown); Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: NL.78977.068.21
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Preoperative; Total Knee Arthroplasty; Prediction; Physical therapy; Physiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients awaiting TKA: Patients awaiting unilateral total knee arthroplasty due to end-stage knee osteoarthritis.
  Interventions: Other: Preoperative assessment

INTERVENTIONS:
Other: Preoperative assessment — Preoperative assessment of physical fitness

SUMMARY:
End-stage KOA results in limitations in activities of daily life (ADL), work and leisure. Treatment for KOA is a stepped care process starting with a conservative approach and in which joint replacement surgery can be considered as the last step. Total knee arthroplasty (TKA) is regarded as the gold standard for the treatment of end-stage knee osteoarthritis (KOA). In 2020, 19.501 TKA surgeries were performed in The Netherlands, end-stage KOA being (97%) the most common reason for surgery.

Until now no risk inventory prediction models have been made for the prediction of physical function at six weeks after TKA. These models may help to distinguish between having a high risk or low risk on a delayed recovery of physical function at six weeks after TKA. This could be beneficial for patients with a high risk. Because than the perioperative process of this patientgroup can be optimized and improved.

DETAILED DESCRIPTION:
Rationale: One of the most common degenerative joint disorders is osteoarthritis (OA). It is most frequently localized in the knee joint. In 2019, the prevalence of knee osteoarthritis (KOA) in the Netherlands reached 704.600 patients. Due to the increase in patients with KOA, healthcare costs are rising. Delayed recovery also causes rising healthcare costs. Preoperative physical fitness turned out to be a predictor of postoperative recovery. A recently published systematic review shows effects of preoperative physical therapy up to 3 months after surgery. To provide therapy to only those who need it, physiotherapeutic care can be optimized and healthcare costs can be saved. Therefore a prediction model, based on physical fitness and patient characteristics, is made to predict the recovery of physical function 6 weeks after total knee arthroplasty.

Objective: To investigate if a risk model can be made, based on physical fitness and patient characteristics, to predict recovery of physical function 6 weeks after total knee arthroplasty. Secondary Objective: To explore if this model is able to distinguish between low risk and high risk of a delayed recovery of physical function.

Study design: Prospective cohort study.

Study population: The study population consists out of patients from the orthopaedic department at the Maastricht University Medical Center + (MUMC+), Zuyderland Medical Centre and the Annadal Clinic, with a diagnosis of end-stage KOA. All patients are scheduled for unilateral primary TKA surgery, because of failing of conservative treatments.

Main study parameters/endpoints: The primary outcome is postoperative physical function (KOOS) 6 weeks after TKA surgery. Predicted by physical fitness and patient characteristics measured during the preoperative assessment. The KOOS is a measurement tool to assess the patients opinion about their knee and associated problems.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: During this examination, the burden on the patient is minimal. The patient will visit the physical therapist once for the preoperative assessment. This appointment will follow already scheduled appointments with the specialist and will last up to 45 minutes. In addition, the subject will receive a one-time phone call. This phone call will be a maximum of 10 minutes, for completing the KOOS questionnaire. The preoperative assessment does not involve any risks.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for primary unilateral TKA surgery
* TKA surgery due to end-stage OA of the knee
* Able to perform the preoperative assessment 4 weeks before surgery
* Able to fulfill the KOOS by phone 6 weeks postoperatively
* Mastery of the Dutch language

Exclusion Criteria:

* Undergoing revision arthroplasty, bilateral TKA or hemi-arthroplasty surgery
* TKA not due to KOA
* Patients who weren't able to perform the preoperative assessment or to fulfill the KOOS postoperatively
* Cognitive impairments
* Complete dependence on a wheelchair
* Unable to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are awaiting unilateral TKA and will be recruited from the orthopeadic departments from the Annadal Clinic, Zuyderland Medical Centre and Maasticht University Medical Center+.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | The KOOS is measured at 6 weeks postoperative
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of the knee injury. The measurement consists out of 42 items, divided in 5 domains (Pain, Symptoms, ADL, leisure and sports and QoL). The total score varies between 0-100. A higher score indicates less knee and knee associated problems.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine F Lenssen, Prof. PhD, Principal Investigator — Maastricht University Medical Center
Locations (3):
- Netherlands (3):
  - Annadal Clinic, Maastricht, Limburg
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Zuyderland Medical Centre, Sittard, Limburg

IPD SHARING:
Plan to Share IPD: No
We do not intent to make IPD available to other researchers.